CLINICAL TRIAL: NCT04625491
Title: Lower Limb Cutaneous Melanoma: Observational Prognostic Study About Specific Location of the Primary Lesion.
Brief Title: Location of Lower Limb Cutaneous Melanomas as a Prognostic Factor.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Antonio Pinero-Madrona, Specialist in Surgery, MD PhD, Hospital Universitario Virgen de la Arrixaca
Other Study IDs: 2020-4-2-HUVA
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cutaneous Melanoma; Anatomical Pathological Condition
Keywords: cutaneous melanoma; lower limb; prognostic
MeSH Terms: conditions — Melanoma; Pathological Conditions, Anatomical | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Location on lower limb: Proximal (thigh) Medium (leg) Distal (ankle and foot)
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
Observational study to know the relevance of specific anatomical location of cutaneous melanoma on lower limbs.

DETAILED DESCRIPTION:
Ambispective (retrospective and prospective) observational register of patients with cutaneous melanoma on lower limbs are grouped in 1) proximal (thigh), 2) medium (leg), and 3) distal (ankle and foot) location. Analysis of melanoma-specific overall and disease-free survival will be made, as well as multivariant analysis for prognostic variables including anatomical location.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous melanoma on the lower limb

Exclusion Criteria:

* Incomplete staging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that were cared of cutaneous melanoma on the lower limb.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Melanoma-specific overall survival | Ten years
  Melanoma-specific overall survival
Melanoma-specific disease-free survival | Ten years
  Melanoma-specific disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Piñero-Madrona, MD PhD, Principal Investigator — Associate Professor of Surgery
Locations (1):
- Hospital Universitario "Virgen de la Arrixaca", Murcia, Spain

IPD SHARING:
Plan to Share IPD: No
An interim analysis of data is planned in 2020.

REFERENCES:
- [Derived] Pinero-Madrona A, Cerezuela-Fuentes P, Ruiz-Merino G, Martinez-Barba E, Ortiz-Reina S, Martinez-Ortiz MJ, Lopez-Avila A, Frias-Iniesta JF, Viney A, Cabezas-Herrera J. Lower limb cutaneous melanoma surgery: location matters. Arch Dermatol Res. 2023 Sep;315(7):1971-1978. doi: 10.1007/s00403-023-02571-z. Epub 2023 Mar 2. PMID 36862181